CLINICAL TRIAL: NCT04596072
Title: A Clinical Trail of Integrative Medicine Approaches for Post-Stroke Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Ruijie Ma, Clinical Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020ZJZS002
Record Dates: First submitted 2020-10-10; First posted 2020-10-22 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Post-stroke Cognitive Impairment
Keywords: post-stroke cognitive impairment; rehabilitation; traditional Chinese medicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): standard treatment
- treatment (Experimental): standard treatment, regular cognitive function training, acupuncture, and herbs
  Interventions: Combination Product: Chinese traditional rehabilitation

INTERVENTIONS:
Combination Product: Chinese traditional rehabilitation — Chinese traditional rehabilitation including acupuncture and herbs
  Arms: treatment

SUMMARY:
The traditional Chinese medicine rehabilitation for the post-stroke cognitive impairment will be intervened, which can promote the recovery of post-stroke cognitive function patients, reduce the disability rate and improve the quality of life.

DETAILED DESCRIPTION:
This study will collect inpatients from April 2019 to December 2024 who from the third affiliated hospital of Zhejiang university of traditional Chinese medicine, Jiaxing hospital of traditional Chinese medicine, Hangzhou hospital of traditional Chinese medicine.this study sets strict time window (stroke recovery, 30-180 days), use multi-center, large sample, randomized controlled study method and the objective recognition rehabilitation evaluation criteria and efficacy evaluation system to evaluate the clinical effect and analysis of health economics.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke as per the TCM definition, presenting symptoms include unilateral paresis or paralysis, sensory deficits, speech impairment, and hemianopsia. PSCI diagnosis involves clinically significant deficits in at least one cognitive domain and severe disruption of instrumental activity of daily livings.
2. age above 18 years;
3. disease duration of 30-180 days;
4. written informed consent by the patient's legal guardian;
5. MoCA (Montreal Cognitive Assessment) score of 17-26. If patient was educated for ≤ 12 years, one score will be deducted;
6. HAMD(Hamilton Depression Scale) score < 20;
7. indications for acupuncture and moxibustion techniques.

Exclusion Criteria:

1. Cognitive impairment caused by subarachnoid hemorrhage, transient ischemic attack, or other intracranial lesions., such as tumors, aneurysms, vascular malformations, cysticercosis, schistosomiasis, encephalitis, meningitis, hydrocephalus, or head trauma;
2. non-atherosclerotic thrombotic cerebral infarction (such as cardiac embolism, procoagulant state, endovascular shedding, or arteritis);
3. pregnant or lactating women;
4. severe chronic diseases of the heart, liver, kidneys, other viscera, or endocrine system or hematopoietic system;
5. severe dementia, serious language understanding disorders, or mental illness;
6. bleeding tendency;
7. lack of inclusion criteria or not suitable for clinical observation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change of Cognitive function | 0 week, 4 weeks, 8 weeks, 12 weeks, 16weeks
  Montreal Cognitive Assessment(MOCA) will be used, this method focus on the sensitivity and specificity of the scale for the recognition of cognitive impairment are high, and it is evaluated from visual spatial/executive function, language function, image ability orientation and so on. MoCA has a maximum score of 30 points. The normal scoring standard is a total score ≥ 26 points (for those with an education level ≤ 12 years, this standard is reduced by 1 point). Higher scores mean a better outcome.

SECONDARY OUTCOMES:
change in the scores of mini-Mental State Examination (MMSE) | 0 week, 8 weeks, 12 weeks, 16 weeks
  The scale is used for rapid evaluation of orientation, memory, attention, calculation, language, and visuospatial structure. MMSE has a maximum score of 30 points. The normal cut-off values are: illiterate group ≥17 points, primary school group ≥20 points, middle school or higher group ≥24 points. Higher scores mean a better outcome.
Changes in Daily Living ability | 0 week, 8 weeks, 12 weeks, 16 weeks
  ADL(Activity of Daily Living) will be used, which also known as the Barthel Index, consists of 10 items, including toileting, grooming, using the toilet, eating, dressing, transferring, activities, going up and down stairs, and bathing). The total score ranges from 0 to 100. Higher scores mean a better outcome.
Changes in depressive status | 0 week, 8 weeks, 12 weeks and 16 weeks
  use Hamilton Depression Scale to evaluate depression, the score were 24 for severe, 17 for moderate and 7 for mild. Higher scores mean a worse outcome.
Changes in the patterns of activation of brain regions related to cognitive impairment | 0 weeks, 8 weeks
  ALLF, fALFF, PerAF, ReHo and DC were used to analyze the resting state functional magnetic resonance imaging. The pattern changes of relevant brain regions related to cognitive impairment after stroke were revealed.

CONTACTS AND LOCATIONS:
Overall Officials: RUIJIE MA, Doctor, Study Director — The Third Affiliated hospital of Zhejiang Chinese Medical University; XINYUN LI, Master, Principal Investigator — Zhejiang Chinese Medical University
Locations (3):
- China (3):
  - The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - Hangzhou hospital of traditional Chinese medicine, Hangzhou, Zhejiang
  - Jiaxing hospital of Chinese traditional medicine, Jiaxing, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided